CLINICAL TRIAL: NCT03794960
Title: A Phase 2b Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of TOL-3021 in Patients With Established Type 1 Diabetes Mellitus
Brief Title: Diabetes AutoimmunitY Withdrawn in Established Patients (DAY)
Acronym: DAY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Modification to Clinical Development Plan
Sponsor: Tolerion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOL-3021-230
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Type 1 Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TOL-3021 (Experimental)
  Interventions: Biological: TOL-3021
- TOL-3021 Placebo (Placebo Comparator)
  Interventions: Other: TOL-3021 Placebo

INTERVENTIONS:
Biological: TOL-3021 — A plasmid expression vector containing the coding sequences for full-length human proinsulin.
  Arms: TOL-3021
Other: TOL-3021 Placebo — TOL-3021 Placebo
  Other Names: Placebo
  Arms: TOL-3021 Placebo

SUMMARY:
The study is a prospective, randomized, double-blind, placebo-controlled, multicenter trial in subjects with established T1D.

DETAILED DESCRIPTION:
The study will include 216 male or female subjects aged 12 to 35 years diagnosed with T1D, as defined by the American Diabetes Association (ADA) criteria and meeting enrollment criteria as follows. Initial enrollment will be restricted to subjects aged 18-35 until an analysis of data from subjects with 3 months' exposure to drug confirms safety. Upon completion of this assessment, enrollment will be open without further restrictions for subjects aged 12-35.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 1 Diabetes Mellitus based on American Diabetes Association (ADA) criteria and within 1.0 to 5.0 years from diagnosis, defined as the first day of insulin administration.
2. Adequate glycemic control for >14 days, defined as 3 consecutive fasting glucose levels by self-administered blood glucose (SMBG) or lab testing <130 mg/dL.
3. Age at randomization of 12.0 - <18.0 years (adolescent), 18.0 - <36.0 years of age (adult) .
4. HbA1c <8.5% based on point-of-care or local lab measurement.

   • Measurement can be repeated every 5-7 days if >8.5%.
5. Presence of antibodies to at least one of the following antigens: GAD-65, IA-2, ZnT8; or insulin.
6. Peak C-peptide during screening 4-hour mixed meal tolerance test (MMTT) ≥ 0.2pmol/mL.
7. Willingness to wear a continuous glucose monitoring (CGM) device for specified periods of time.
8. Written informed consent, including authorization to release health information and assent for adolescent subjects.
9. Willingness and ability of subject or adult guardian to comply with all study procedures of the study protocol, including attending all clinic visits.

Exclusion Criteria:

1. Body Mass Index (BMI) >30 kg/m2 for adults; >95 percentile BMI-for-age for subjects under 18 years of age.
2. Previous immunotherapy for T1D.
3. Diagnosis of liver disease or hepatic enzymes, as defined by ALT and/or AST ≥ 2.5 times the upper limit of normal (ULN).
4. Hematology: white blood cells (WBC) <3 x 109/L; platelets <100 x 109/L; hemoglobin <10.0 g/dL. (Low WBC values may be repeated every 3-7 days, and results to be discussed with the Medical Monitor.)
5. Serum creatinine >1.5 times ULN.
6. History of malignancy, except for cancers in remission >5 years, or basal cell or in situ squamous cell carcinoma of the skin.
7. Significant cardiovascular disease (including inadequately controlled hypertension), history of myocardial infarction, angina, use of anti-anginal medicines (e.g., nitroglycerin), or abnormal stress test, which, in the opinion of the Principal Investigator (PI), would interfere with participation in the trial.
8. Immunosuppressive therapy (systemic corticosteroids, cyclosporine, azathioprine, or biologics) within 30 days of screening.
9. Current or prior (within the last 30 days) use of metformin, sulfonylureas, glinides, thiazolidinediones, GLP1-RAs, DPP-IV inhibitors, pramlintide, or SGLT-2 inhibitors.
10. Current use of verapamil or α-methyldopa.
11. History of any organ transplant, including islet cell transplant.
12. Active autoimmune or immune deficiency disorder other than T1D or well-controlled autoimmune thyroid disease (e.g., sarcoidosis, rheumatoid arthritis, moderate-to-severe psoriasis, inflammatory bowel disease, and other autoimmune conditions that may require treatment with TNF or other biologics), unless approved by the Medical Monitor.
13. Thyroid-stimulating hormone (TSH) at screening >2.5 mIU/L.
14. History of adrenal insufficiency.
15. Evidence of infection with HBV (as defined by hepatitis B surface antigen, HBsAg), HCV (anti-HCV antibodies), or HIV.
16. Positive urine pregnancy test: Females of childbearing potential must be excluded if they have a positive urine pregnancy test at screening or randomization or if they are not using medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, IUD, progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or 1 year or more postmenopausal must be specified in the subject's Case Report Form (CRF).
17. Males of reproductive potential who are unwilling to use medically acceptable birth control, unless the female partner is postmenopausal or surgically sterile.
18. Any social condition or medical condition that would, in the opinion of the PI, prevent complete participation in the study or would pose a significant hazard to the subject's participation.
19. Anticipated major surgery during the duration of the trial, which could interfere with participation in the trial.
20. History of drug or alcohol dependence within 12 months of screening.
21. Psychiatric disorder that would prevent subjects from giving informed consent.
22. Participation in other studies involving the administration of an investigational drug or device, including the administration of an experimental agent for T1D, at any time, or use of an experimental device for T1D within 30 days prior to screening, unless approved by the Medical Monitor.

Ages: 12 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-14 (Estimated); Primary Completion 2021-12-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Treatment Effect | at Week 52
  The primary outcome is the treatment effect on log-transformed MMTT C-peptide area under the curve (AUC) after 52 weeks of TOL-3021 treatment

SECONDARY OUTCOMES:
Rate of Clinically important hypoglycemia as defined by measured glucose value of <54 mg/dL (3.0 mM/L) | at Week 52
  By glucometer, a single blood glucose level
Rate of Clinically important hypoglycemia as defined by measured glucose value of <54 mg/dL (3.0 mM/L) | at Week 52
  By CGM, ≥15 consecutive minutes with glucose <54 mg/dL
Rate of Clinically important hypoglycemia as defined by measured glucose value of <54 mg/dL (3.0 mM/L) | at Week 52
  Total daily insulin requirements in units per kilogram (kg) body weight
Rate of Clinically important hypoglycemia as defined by measured glucose value of <54 mg/dL (3.0 mM/L) | at Week 52
  HbA1c
Clinical responder analysis | at Week 52
  Proportion of subjects in each treatment arm with HbA1c levels less than 6.5% at Week 52
Clinical responder analysis | at Week 52
  Measure by GMS - Time in range 70 - 80 mg/dL
Clinical responder analysis | at Week 52
  Measure by GMS - Time >180 mg/dL
Clinical responder analysis | at Week 52
  Measure by GMS - Time >250 mg/dL
Clinical responder analysis | at Week 52
  Measure by GMS - Mean Glucose Coefficient of Variation
Clinical responder analysis | at Week 52
  Measure by GMS - Low Blood Glucose Index (LBGI)
Clinical responder analysis | at Week 52
  Measure by GMS - Glucose below 70 mg/dL Area Over the Curve (AOC70)
Other measures of hypoglycemia | at Week 52
  Severe hypoglycemia (SH) events (impaired or loss of consciousness requiring assistance of another)
Other measures of hypoglycemia | at Week 52
  Documented symptomatic hypoglycemia (an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <70 mg/dl (3.9 mmol/L))
Other measures of hypoglycemia | at Week 52
  Total time <70 mg/dL by CGM
Other measures of hypoglycemia | at Week 52
  Nocturnal hypoglycemia, severe or documented symptomatic episodes (as defined above) occurring after the subject has retired for the primary sleeping period
Immunologic | at Week 52
  Quantum dot (Q-dot) responses within the qualifying subpopulation to confirm induction of specific autoantigen tolerance
Immunologic | at Week 52
  Comparison of quantum dot responses within the qualifying subpopulation to clinical outcomes to confirm correlation with specific autoantigen tolerance.
Immunologic | at Week 52
  Determine effect of treatment on and predictive value of regulatory/protective humoral immune response to proinsulin/insulin
Immunologic | at Week 52
  Determine effect of treatment on and predictive value of serum insulin autoantibody affinity for subjects
Immunologic | at Week 52
  Determine effect of treatment on and predictive value of Insulin autoantibody isotypes (IgA and IgM) and IgG subclasses
Immunologic | at Week 52
  Determine effect of treatment on and predictive value of serum insulin, glutamic acid decarboxylase, IA-2, and ZnT8 antibodies by highly sensitive ECL assay
Immunologic | at Week 52
  Determine effect of treatment on and predictive value of competition assays of serum insulin and proinsulin IgM and IgG antibodies

IPD SHARING:
Plan to Share IPD: Undecided